CLINICAL TRIAL: NCT03952611
Title: Three Arm Prospective Randomized Controlled Trial of HD White-light Colonoscopy vs HD White-light Colonoscopy With Reveal® Distal Attachment Cap Versus HD White-light Colonoscopy With Endocuff Vision for the Detection of Colorectal Adenomas
Brief Title: Three Arm Rand Trial of HD Light vs Reveal® Cap vs Endocuff Cap for Detection of Colorectal Adenomas (TRACE)
Acronym: TRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Biomedical Research Foundation (Other)
Responsible Party: Sponsor
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: RND#00978
Record Dates: First submitted 2017-10-23; First posted 2019-05-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Adenoma
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: Three Arm Randomized Control Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization will be done by computer allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- High-Definition White-light Colonoscopy (Active Comparator): Using an instrument called colonoscope which is used to detect colonic polyps
  Interventions: Procedure: Colonoscopy
- High-Definition White-light Colonoscopy With Reveal® (Active Comparator): Using an instrument called cap at end of colonoscope which is used to straighten colon folds
  Interventions: Procedure: Colonoscopy; Device: distal Cap
- High-Definition White-light Colonoscopy With Endocuff Vision (Active Comparator): Using an instrument called Endocuff at end of colonoscope which is used to straighten colon folds
  Interventions: Procedure: Colonoscopy; Device: Endocuff

INTERVENTIONS:
Procedure: Colonoscopy — Using an instrument called colonoscope which is used to detect colonic polyps
Device: distal Cap — Using an instrument called cap at end of colonoscope which is used to straighten colon folds
  Arms: High-Definition White-light Colonoscopy With Reveal®
Device: Endocuff — Using an instrument called Endocuff at end of colonoscope which is used to straighten colon folds
  Arms: High-Definition White-light Colonoscopy With Endocuff Vision

SUMMARY:
Protocol Title: Three Arm Prospective Randomized controlled trial of High-Definition White-light colonoscopy versus High-Definition White-light colonoscopy with Reveal® Distal Attachment Cap versus High-Definition White-light colonoscopy with Endocuff Vision for the detection of colorectal adenomas

Hypothesis: Detection rate of adenomas in patients will be higher in procedures performed with High-Definition White-light (HDWL) colonoscopy with Reveal® distal attachment cap and HDWL colonoscopy with Endocuff Vision compared to HDWL colonoscopes alone

Design: Multicenter, Prospective, randomized controlled study

Primary Aim: To compare the proportion of subjects with at least one adenoma detected during HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.

Secondary Aims: To compare the number of adenomas detected per subject with HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.

To compare the detection rates for polyp subtypes (including advanced adenomas, serrated polyps, right sided adenomas, etc.), cecal intubation rate, insertion time, withdrawal time, and complications of HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.

DETAILED DESCRIPTION:
Hypothesis and specific aims of the Study

We hypothesize that the detection rate of patients with colorectal adenomas will be higher with HDWL colonoscopy with Reveal® distal attachment cap and HDWL colonoscopy with Endocuff Vision compared to HDWL colonoscopy alone.

Primary Aim:

To compare the proportion of subjects with at least one adenoma detected during HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.

Secondary Aims:

1. To compare the number of adenomas detected per subject with HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.
2. To compare the detection rates for polyp subtypes (including advanced adenomas, serrated polyps, right sided adenomas, etc.), cecal intubation rate, insertion time, withdrawal time, and complications of HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.

Methodology:

This will be a prospective, randomized controlled study. Subjects referred for screening or surveillance colonoscopy will be prospectively enrolled. They will be randomized to one of 3 arms, i.e. HDWL colonoscopy HDWL colonoscopy with Reveal® cap or HDWL colonoscopy with Endocuff Vision.

Enrollment:

A member of the research team will approach a potential subject to discuss participation in the study, including background of the proposed study, inclusion and exclusion criteria, benefits and risks of the procedures and follow-up. If this is of interest to the subject, the informed consent form is discussed and presented. The subject must sign the consent form prior to enrollment. This form will have prior approval of the study site's Institutional Review Board (IRB). Failure to obtain informed consent renders the subject ineligible for the study.

Length of the study:

The duration of the study is expected to be approximately 12 months. Enrollment of study patients will cease when approximately 1227 patients have been enrolled.

Inclusion criteria

* Referral for screening or surveillance colonoscopy
* Ability to provide informed consent

Exclusion criteria

* Prior history of colon cancer
* History of inflammatory bowel disease
* Prior surgical resection of any part of the colon
* Use of anti-platelet agents or anticoagulants that precludes the removal of polyps during the procedure
* History of polyposis syndrome or HNPCC
* Inability to give informed consent
* Family history of colon cancer in a first degree relative < 60 years or two first degree relatives with colorectal cancer

For three groups, moderate sedation will be administered in a standard fashion with intravenous midazolam, meperidine or fentanyl prior to undergoing colonoscopy.

The colonoscope (HDWL colonoscope or HDWL colonoscope with Reveal® cap or HDWL colonoscope with Endocuff Vision) will be inserted and cecum will be intubated. Photo documentation of the cecum will be performed. The colonic mucosa will be carefully visualized upon withdrawal of the colonoscope.

The time from the point of insertion of the colonoscope into the rectum to the intubation of cecum will be recorded with a stop watch by a research coordinator and will be documented as the "insertion time".

The time spent in inspecting the mucosa during withdrawal of the colonoscope will be documented as the "withdrawal time". During withdrawal of the colonoscope the stop watch will be stopped whenever mucosa is being cleaned, fluid/solid debris is suctioned or a polyp is being removed to ensure that the withdrawal time is the actual representation of the mucosal inspection time. Meticulous technique will be employed during the withdrawal phase with special efforts to visualize portions of colonic mucosa on the proximal aspects of haustral folds, flexures and valves.

All polyps detected will be documented: size, location, and morphology (using the Paris classification - Appendix A). Photo documentation of the polyps will be performed.

Polyps will then be removed with a biopsy forceps or snare and sent for histopathological evaluation, each in a separate jar and labeled accordingly.

The bowel preparation will be evaluated and graded according to previously reported criteria using the Boston Bowel Preparation Scale (Appendix B). Complications including any mucosal trauma from the high definition colonoscope alone or with high definition colonoscope with Reveal® cap or Endocuff Vision, perforation or gastrointestinal bleeding (requiring intervention) will be recorded for three groups.

ELIGIBILITY:
Inclusion Criteria:

* Referral for screening or surveillance colonoscopy
* Ability to provide informed consent

Exclusion Criteria:

* Prior history of colon cancer
* History of inflammatory bowel disease
* Prior surgical resection of any part of the colon
* Use of anti-platelet agents or anticoagulants that precludes the removal of polyps during the procedure
* History of polyposis syndrome or HNPCC
* Inability to give informed consent
* Family history of colon cancer in a first degree relative < 60 years or two first degree relatives with colorectal cancer

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1203 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | Through the study (1 year)
  To compare the proportion of subjects with at least one adenoma detected during HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.

SECONDARY OUTCOMES:
Number of Adenomas per person | Through the study (1 year)
  To compare the number of adenomas detected per subject with HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.
detection rates of advanced adenomas | Through the study (1 year)
  To compare the detection rates for advanced adenomas of HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.
detect rates of serrated polyps | Through the study (1 year)
  To compare the detection rates for serrated polyps of HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.
detect rates of right sided adenomas | Through the study (1 year)
  To compare the detection rates of right sided adenomas of HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.
to determine cecal intubation time | Through the study (1 year)
  To compare the cecal intubation time of HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.
to determine insertion and withdrawal time | Through the study (1 year)
  To compare the insertion and withdrawal time of the procedure of HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.
to determine complications | Through the study(1 year)
  To compare the complications of procedure of HDWL colonoscopy versus HDWL colonoscopy with Reveal® distal attachment cap versus HDWL colonoscopy with Endocuff Vision.

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Kansas City VA Hospital
Locations (1):
- Kansas City VA Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This is a multi- center study and we will receive de identified data from other centered via REDCAP

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Background] Winawer SJ, Zauber AG, Fletcher RH, Stillman JS, O'Brien MJ, Levin B, Smith RA, Lieberman DA, Burt RW, Levin TR, Bond JH, Brooks D, Byers T, Hyman N, Kirk L, Thorson A, Simmang C, Johnson D, Rex DK; US Multi-Society Task Force on Colorectal Cancer; American Cancer Society. Guidelines for colonoscopy surveillance after polypectomy: a consensus update by the US Multi-Society Task Force on Colorectal Cancer and the American Cancer Society. Gastroenterology. 2006 May;130(6):1872-85. doi: 10.1053/j.gastro.2006.03.012. PMID 16697750
- [Background] Citarda F, Tomaselli G, Capocaccia R, Barcherini S, Crespi M; Italian Multicentre Study Group. Efficacy in standard clinical practice of colonoscopic polypectomy in reducing colorectal cancer incidence. Gut. 2001 Jun;48(6):812-5. doi: 10.1136/gut.48.6.812. PMID 11358901
- [Background] van Rijn JC, Reitsma JB, Stoker J, Bossuyt PM, van Deventer SJ, Dekker E. Polyp miss rate determined by tandem colonoscopy: a systematic review. Am J Gastroenterol. 2006 Feb;101(2):343-50. doi: 10.1111/j.1572-0241.2006.00390.x. PMID 16454841
- [Background] Heresbach D, Barrioz T, Lapalus MG, Coumaros D, Bauret P, Potier P, Sautereau D, Boustiere C, Grimaud JC, Barthelemy C, See J, Serraj I, D'Halluin PN, Branger B, Ponchon T. Miss rate for colorectal neoplastic polyps: a prospective multicenter study of back-to-back video colonoscopies. Endoscopy. 2008 Apr;40(4):284-90. doi: 10.1055/s-2007-995618. PMID 18389446
- [Background] Floer M, Biecker E, Fitzlaff R, Roming H, Ameis D, Heinecke A, Kunsch S, Ellenrieder V, Strobel P, Schepke M, Meister T. Higher adenoma detection rates with endocuff-assisted colonoscopy - a randomized controlled multicenter trial. PLoS One. 2014 Dec 3;9(12):e114267. doi: 10.1371/journal.pone.0114267. eCollection 2014. PMID 25470133
- [Background] Rastogi A, Bansal A, Rao DS, Gupta N, Wani SB, Shipe T, Gaddam S, Singh V, Sharma P. Higher adenoma detection rates with cap-assisted colonoscopy: a randomised controlled trial. Gut. 2012 Mar;61(3):402-8. doi: 10.1136/gutjnl-2011-300187. Epub 2011 Oct 13. PMID 21997547
- [Background] Biecker E, Floer M, Heinecke A, Strobel P, Bohme R, Schepke M, Meister T. Novel endocuff-assisted colonoscopy significantly increases the polyp detection rate: a randomized controlled trial. J Clin Gastroenterol. 2015 May-Jun;49(5):413-8. doi: 10.1097/MCG.0000000000000166. PMID 24921209
- [Derived] Desai M, Rex DK, Bohm ME, Davitkov P, DeWitt JM, Fischer M, Faulx G, Heath R, Imler TD, James-Stevenson TN, Kahi CJ, Kessler WR, Kohli DR, McHenry L, Rai T, Rogers NA, Sagi SV, Sathyamurthy A, Vennalaganti P, Sundaram S, Patel H, Higbee A, Kennedy K, Lahr R, Stojadinovikj G, Campbell C, Dasari C, Parasa S, Faulx A, Sharma P. Impact of withdrawal time on adenoma detection rate: results from a prospective multicenter trial. Gastrointest Endosc. 2023 Mar;97(3):537-543.e2. doi: 10.1016/j.gie.2022.09.031. Epub 2022 Oct 10. PMID 36228700
- [Derived] Desai M, Rex DK, Bohm ME, Davitkov P, DeWitt JM, Fischer M, Faulx G, Heath R, Imler TD, James-Stevenson TN, Kahi CJ, Kessler WR, Kohli DR, McHenry L, Rai T, Rogers NA, Sagi SV, Sathyamurthy A, Vennalaganti P, Sundaram S, Patel H, Higbee A, Kennedy K, Lahr R, Stojadinovikj G, Dasari C, Parasa S, Faulx A, Sharma P. High-Definition Colonoscopy Compared With Cuff- and Cap-Assisted Colonoscopy: Results From a Multicenter, Prospective, Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2022 Sep;20(9):2023-2031.e6. doi: 10.1016/j.cgh.2021.12.037. Epub 2021 Dec 31. PMID 34979245